CLINICAL TRIAL: NCT00502775
Title: A Comparison of Fluticasone Furoate Nasal Spray Versus Oral Fexofenadine in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Fluticasone Furoate Nasal Spray Versus Oral Fexofenadine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFU109047
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2009-03-20 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: ragweed; once daily; fexofenadine; fluticasone furoate; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — fluticasone furoate; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluticasone furoate, fexofenadine
  Other Names: fluticasone furoate; fexofenadine

SUMMARY:
The primary objective of the study is to compare nighttime symptom relief of fluticasone furoate nasal spray versus oral fexofenadine

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Otherwise healthy outpatient with mountain cedar allergy
* Male or eligible female Females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control
* Age 12 years or older at Visit 2
* Diagnosis of seasonal allergic rhinitis (SAR) to mountain cedar
* Adequate exposure to mountain cedar pollen
* Ability to comply with study procedures
* Literate

Exclusion criteria:

* Significant concomitant medical conditions
* Use of intranasal corticosteroids within four weeks prior to Visit 1; use of inhaled, oral, intramuscular, intravenous, ocular, and/or dermatological corticosteroid (with the exception of hydrocortisone cream/ointment, 1% or less) within eight weeks prior to Visit 1.
* Use of other allergy medications within specific timeframes relative to Visit 1
* Use of other medications that may affect allergic rhinitis or its symptoms
* Use of immunosuppressive medications eight weeks prior to screening and during the study
* Immunotherapy patients who are not stable on current dose
* Use of any medications that significantly alters the pharmacokinetics of fluticasone furoate or fexofenadine
* Allergy/Intolerance to corticosteroids, antihistamines, or any excipients in the two products
* Use of contact lenses
* Recent clinical trial/experimental medication experience within 30 days of Visit 1
* Subject previously failed the 21-day screen period or failed to complete the treatment period
* Positive or inconclusive pregnancy test or female who is breastfeeding
* Employee or relative affiliation with investigational site
* Current tobacco use
* Active chickenpox or measles or exposure in the last 3 weeks

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (40):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFU109047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Started | 229 | 224 | 227
Completed | 219 | 209 | 214
Not Completed | 10 | 15 | 13
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Protocol Violation | 1 | 5 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Sponsor Terminated Study | 1 | 0 | 1
Not completed — Non-compliance with eDiary | 4 | 1 | 1
Not completed — Subject unable to swallow capsule | 1 | 0 | 1
Not completed — Logpad compliance <80% | 1 | 0 | 0
Not completed — Randomized in error | 0 | 1 | 1
Not completed — Non-compliance | 0 | 2 | 2
Not completed — Outside pollen area more than 48 hours | 0 | 1 | 0
Not completed — Declining pollen counts | 0 | 1 | 1
Not completed — Subject in jail | 0 | 1 | 0
Not completed — Subject took disallowed drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg | Total
Number analyzed (Participants) | 229 | 224 | 227 | 680
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (12.71) | 34.0 (13.55) | 34.3 (13.66) | 34.4 (13.29)
Gender [Count of Participants; unit: Participants]
  Female | 139 | 152 | 135 | 426
  Male | 90 | 72 | 92 | 254
Race/Ethnicity, Customized [Number; unit: Number of Participants]
  White | 181 | 189 | 181 | 551
  African American | 40 | 29 | 42 | 111
  Other | 8 | 6 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Nighttime Symptom Score (NSS)
Description: Questions include: 1. Nasal congestion on awakening (Score: 0=none, 1=mild, 2=moderate, 3=severe); 2. Difficulty going to sleep (Score: 0=not at all, 1=little, 2=moderately, 3=very); 3. Nighttime awakenings (Score: 0=not at all, 1=once, 2=more than once, 3=felt like awake all night). The sum of the ratings for the three items comprises the NSS.
Time Frame: Baseline and Weeks 1-2
Population: One analysis population was defined for this study, the Intent-to-Treat population. . The Intent-to-Treat (ITT) population included all subjects randomized to double-blind treatment. This population formed the basis for all summaries of demographic, background, efficacy, and safety data.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.3 (0.11) | -3.1 (0.12) | -2.2 (0.12)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110mcg vs Fexofenadine 180 mg; The primary efficacy measure, mean change from baseline over the two-week treatment period in NSS compared between fluticasone furoate and fexofenadine, was assessed at a significance level of α=0.05. If the null hypothesis of this comparison was rejected, then the secondary measures were subject to hypothesis testing. The study was powered at 90%; Test type: Superiority or Other; p < 0.001, ANCOVA — Symptom scores were grouped in 3 families: nasal, ocular, instantaneous. Within each family, results of hypothesis tests were adjusted using Hochberg's method; No other strata or covariates, other than investigator, were defined; Mean Difference (Net) = -0.9, 95% CI [-1.2 to -0.6], Standard Error of Mean 0.16 — Mean Difference = Mean Change in Fluticasone Furoate - Mean Change in Fexofenadine
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 110mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.8, 95% CI [-1.1 to -0.4], Standard Error of Mean 0.16 — Mean Difference = Mean Change in Fluticasone Furoate - Mean Change in Placebo
Statistical Analysis 3: Comparison: Placebo vs Fexofenadine 180 mg; Test type: Superiority or Other; p = 0.374, ANCOVA; Mean Difference (Net) = 0.1, 95% CI [-0.2 to 0.5], Standard Error of Mean 0.16 — Mean Difference = Mean Change in Fexofenadine - Mean Change in Placebo

2. Secondary Outcome: Mean Change From Baseline in Nighttime Reflective Total Nasal Symptom Score (N-rTNSS)
Description: Subjects assessed four nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing). The sum of the four nasal symptoms comprised the total nasal symptom score (TNSS). Reflective rating represented symptoms over preceding 12 hours. Scores: 0=symptoms not present, 1=mild severity, 2=moderate severity, 3=severe.
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.9 (0.15) | -4.1 (0.17) | -2.9 (0.16)

3. Secondary Outcome: Mean Change From Baseline in Daytime Reflective Total Nasal Symptom Score (D-rTNSS)
Description: as for outcome 2
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -3.0 (0.15) | -4.2 (0.18) | -2.9 (0.16)

4. Secondary Outcome: Mean Change From Baseline in 24 Hour Reflective Total Nasal Symptom Score (24 Hour rTNSS)
Description: Subjects assessed four nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing). The sum of the four nasal symptoms comprised the total nasal symptom score (TNSS).Reflective rating represented symptoms over preceding 12 hours. Scores: 0=symptoms not present, 1=mild severity, 2=moderate severity, 3=severe.
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.8 (0.14) | -4.1 (0.18) | -2.8 (0.16)

5. Secondary Outcome: Mean Change From Baseline in Nighttime Reflective Total Ocular Symptom Score (N-rTOSS)
Description: Subjects assessed three ocular symptoms (itching/ burning eyes, tearing/watering eyes, and eye redness). The sum of the 3 ocular symptoms comprised the total ocular symptom score (TOSS). Reflective rating represented symptoms over preceding 12 hours. Scores: 0=symptoms not present, 1=mild severity, 2=moderate severity, 3=severe.
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.3 (0.13) | -2.7 (0.14) | -2.2 (0.13)

6. Secondary Outcome: Mean Change From Baseline in Daytime Reflective Total Ocular Symptom Score (D-rTOSS)
Description: as for outcome 5
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.5 (0.13) | -2.9 (0.14) | -2.4 (0.13)

7. Secondary Outcome: Mean Change From Baseline in 24 Hour Reflective Total Ocular Symptoms Score (rTOSS)
Description: as for outcome 5
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.3 (0.13) | -2.7 (0.14) | -2.2 (0.13)

8. Secondary Outcome: Mean Change From Baseline in Pre-Dose Instantaneous Total Nasal Symptom Score (iTNSS)
Description: Subjects assessed four nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing). The sum of the four nasal symptoms comprised the total nasal symptom score (TNSS).Instantaneous rating represented symptoms at the time of the assessment. Scores: 0=symptoms not present, 1=mild severity, 2=moderate severity, 3=severe.
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.8 (0.15) | -4.1 (0.18) | -2.7 (0.17)

9. Secondary Outcome: Mean Change From Baseline in Pre-Dose Instantaneous Total Ocular Symptom Score (iTOSS)
Description: Subjects assessed three ocular symptoms (itching/ burning eyes, tearing/watering eyes, and eye redness). The sum of the four ocular symptoms comprised the total nasal symptom score (TOSS).Instantaneous rating represented symptoms at the time of the assessment. Scores: 0=symptoms not present, 1=mild severity, 2=moderate severity, 3=severe.
Time Frame: Baseline and Weeks 1-2
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 228 | 224 | 226
Score on a Scale | -2.2 (0.13) | -2.7 (0.14) | -2.2 (0.14)

10. Secondary Outcome: Mean Change From Baseline in Morning Peak Nasal Inspiratory Flow (PNIF)
Description: Subjects used a portable hand-held inspiratory flow meter to measure and record PNIF in the morning prior to taking the study medication. Three measurements were taken and the highest measurement was recorded in the electronic diary. A positive change signifies improved nasal air flow.
Time Frame: Baseline and Weeks 1-2
Population: Two subjects in the placebo group & three in the FFNS group recorded no data during the two-week treatment period.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 226 | 221 | 226
Score on a Scale | 4.8 (1.27) | 13.0 (1.61) | 2.2 (1.21)

11. Secondary Outcome: Mean Change From Baseline in Evening Peak Nasal Inspiratory Flow (PNIF)
Description: Subjects used a portable hand-held inspiratory flow meter to measure and record PNIF in the evening. Three measurements were taken and the highest measurement was recorded in the electronic diary. A positive change signifies improved nasal air flow.
Time Frame: Baseline and Weeks 1-2
Population: Two subjects in the placebo group & two in the FFNS group recorded no data during the two-week treatment period.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 226 | 222 | 226
Score on a Scale | 2.3 (1.38) | 9.7 (1.73) | 0.3 (1.37)

12. Secondary Outcome: Mean Change From Baseline at Day 15 for Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ)
Description: Subjects completed the 16-item Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ)to assess nocturnal rhinitis-related quality of life. The NRQLQ measures the functional problems most troublesome to patients with nocturnal allergy symptoms. Each question scored from 0-6 with higher scores indicating more nocturnal impairment.
Time Frame: Baseline, Day 15 or if Early Withdrawal Day
Population: Ten placebo subjects, six FFNS subjects, and four fexofenadine subjects had no overall NRQLQ score at endpoint, indicating either a missing score for one or more of the NRQLQ domains, a missing baseline score, or both. One additional FFNS patient had no on-treatment NRQLQ data.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Number analyzed (Participants) | 218 | 217 | 222
Score on a Scale | -1.4 (0.09) | -2.0 (0.10) | -1.4 (0.10)

ADVERSE EVENTS:
Arm/Group | Placebo | Fluticasone Furoate 110mcg | Fexofenadine 180 mg
Serious Adverse Events (participants affected / at risk) | 0/229 | 0/224 | 1/227
Other Adverse Events (participants affected / at risk) | 27/229 | 31/224 | 37/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=229) | Fluticasone Furoate 110mcg (N=224) | Fexofenadine 180 mg (N=227)
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=229) | Fluticasone Furoate 110mcg (N=224) | Fexofenadine 180 mg (N=227)
Headache (Nervous system disorders) | 6 | 10 | 9
Sinus headache (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Human bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1
Feeling jittery (General disorders) | 0 | 1 | 0
Ill-defined disorder (General disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.